CLINICAL TRIAL: NCT00956553
Title: A Phase IV, Randomised Study to Evaluate the Immune Responses of UK Adolescent Girls Receiving CervarixTM or GardasilTM Human Papillomavirus Vaccines
Brief Title: Reactogenicity Study of Cervarix and Gardasil in UK Adolescent Girls
Acronym: HPV CSP01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPV CSP01
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2018-08

CONDITIONS: HPV Infections
Keywords: HPV; Human Papilloma Virus; Cervical cancer vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervarix (Active Comparator): Three doses of Cervarix at month 0, 1 and 6. Blood sample at month 0, 2, 7 and 12. Optional vaginal sponge sample at month 7.
  Interventions: Biological: Cervarix
- Gardasil (Active Comparator): Three doses of Gardasil at month 0, 1 and 6. Blood sample at month 0, 2, 7 and 12. Optional vaginal sponge sample at month 7.
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: Cervarix — Three doses of Cervarix at month 0, 1 and 6.
  Arms: Cervarix
Biological: Gardasil — Three doses of Gardasil at month 0, 1 and 6.
  Arms: Gardasil

SUMMARY:
This is a phase IV study to evaluate the body's immune response of participants to the Cervarix and Gardasil vaccines against the Human Papilloma Virus (HPV) types associated with increased risk of cervical cancer.

DETAILED DESCRIPTION:
This study looks at possible cross reactivity between different HPV serotypes and both peripheral antibodies and mucosally-secreted antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 13 and 15 years at the time of the first immunisation
* Female
* No contraindications to vaccination as specified in the "Green Book" - Immunisation Against Infectious Disease, HMSO.
* Written informed consent obtained from parent or guardian of subject

Exclusion Criteria:

* Pregnant or become pregnant during the course of the trial (no contraindications to vaccination for those taking the contraceptive pill).
* Breast-feeding mothers
* Allergic to vaccine components

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Measurable antibody mediated neutralisation of HPV serotype 6, 11, 16, 18 and genetically related serotypes, especially 45 | 18 months from enrollment

SECONDARY OUTCOMES:
Determine differences in vaccine formulation and their impact on cross protection. | 24 months from enrollment

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Public Health England, Stevenage, Hertfordshire
  - Professor Elizabeth Miller, Gloucester
  - Public Health England, London

REFERENCES:
- [Result] Haskins-Coulter T, Southern J, Andrews N, Miller E. Reactogenicity of Cervarix and Gardasil human papillomavirus (HPV) vaccines in a randomized single blind trial in healthy UK adolescent females. Hum Vaccin Immunother. 2017 Jun 3;13(6):1-9. doi: 10.1080/21645515.2016.1277846. Epub 2017 Mar 20. PMID 28319456
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Godi A, Panwar K, Haque M, Cocuzza CE, Andrews N, Southern J, Turner P, Miller E, Beddows S. Durability of the neutralizing antibody response to vaccine and non-vaccine HPV types 7 years following immunization with either Cervarix(R) or Gardasil(R) vaccine. Vaccine. 2019 Apr 24;37(18):2455-2462. doi: 10.1016/j.vaccine.2019.03.052. Epub 2019 Mar 27. PMID 30926298
- [Derived] Draper E, Bissett SL, Howell-Jones R, Waight P, Soldan K, Jit M, Andrews N, Miller E, Beddows S. A randomized, observer-blinded immunogenicity trial of Cervarix((R)) and Gardasil((R)) Human Papillomavirus vaccines in 12-15 year old girls. PLoS One. 2013 May 1;8(5):e61825. doi: 10.1371/journal.pone.0061825. Print 2013. PMID 23650505
- See also: Published study results — https://www.ncbi.nlm.nih.gov/pubmed/28319456